CLINICAL TRIAL: NCT03893305
Title: Pattern of Skin Disorders in Geriatric Population
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Rizk Melad, residant, Assiut University
Other Study IDs: skin disorders in geriatric
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Geriatric Skin Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators attempt to determine the frequency of dermatologic diseases in geriatric patients, and search for seasonal, age-related, gender-related and socio- demographic differences in geriatric patients attending the outpatient clinic of the Department of Dermatology, Venereology and Andrology in Assiut University Hospital.

DETAILED DESCRIPTION:
Geriatric health care has become a worldwide concern, but relatively few statistical studies are available about geriatric skin diseases (liao et al., 2001). There are published studies regarding skin disorders among the elderly population from different countries such as Taiwan, USA, Norway, the Philippines and Turkey (Mcfadden and Hande 1989). All of these studies are about detecting the prevalence or characteristic pattern of skin diseases, or identifying past or present skin complaints and the dermatologic findings in the elderly (Tianco et al.,1992).

Although there is no exact age for getting old, 65 years is usually accepted as the beginning (Blackman et al., 1999). However, life expectancy is increasing all over the world and the geriatric population is rising dramatically every year as the medical care improves (Beek and Jones, 2000). Aging is a complex multifactorial phenomenon in which progressive intrinsic changes in the skin combine synergistically with cumulative environment insults to produce both structural and functional disturbances (Beauregard and Gilchrest, 1987).

Two types of skin aging exist, which may be divided into intrinsic aging, which includes those changes that are due to normal maturity and occur in all individuals, and extrinsic aging, produced by extrinsic factors such as ultraviolet light exposure, smoking, and environmental pollutants (Norman, 2001). Better understanding of the underlying mechanisms accompanying skin aging could constitute the basis for extending the lifespan in good health (American Geriatrics Society 2015).

The frequencies of some diseases change with advancing age. Incidence of eczematous dermatitis gradually decreases with age, may be due to more contact with environmental and physical factors (Havlik et al., 1999).

Population with old aged skin show a decline in the regular functions of skin, including cell replacement capacity, wound healing, immune responsiveness, decline in appendegeal functions and DNA repair capacity which may be responsible for the higher incidence of sun-related diseases and cutaneous malignancies in elderly people. (Yaar and Gilchrest, 1999).

Pruritic skin diseases are the most common dermatological problem in the elderly. Pruritis can be psychogenic in origin. However, there are a number of dermatological and metabolic conditions that involve pruritis. Xerosis is the most common underlying dermatological condition. (Norman, 2003) Decreased mobility, drug-induced disorders, and increased incidences of many chronic diseases are among the reasons elderly individuals are at heightened risk for skin diseases. Atherosclerosis, diabetes mellitus, human immunodeficiency virus (HIV), and congestive heart failure are some disease processes that can be detrimental to skin. These diseases are known to impede vascular efficiency and decrease immune responses, thereby reducing the body's ability to heal (Norman, 2001).

Decreased immune surveillance in the elderly provides more opportunity for the development of bacterial and viral infections in these patients (Elgart, 2002).

Decreases in personal care, epidermal turnover, and immunologic functions are observed, possibly responsible for the high prevalence of fungal infections (Havlik et al., 1999).

ELIGIBILITY:
Inclusion Criteria:

* All Patients aged 65 years and older

Exclusion Criteria:

* No exclusion criteria

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: • Patients aged 65 years and older attending to the dermatology outpatient clinics over a forward one year period (as an antegrade study) and another six year retrograde
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
determine the frequency of dermatologic diseases in geriatric patients | seven years
  search for seasonal, age-related, gender-related and socio- demographic differences in geriatric patients

CONTACTS AND LOCATIONS:
Overall Officials: Reham M Abdel Gaber, Lecture, Study Director — Supervisor
Locations (1):
- Kerolos R.Melad, Asyut, Egypt